CLINICAL TRIAL: NCT06188104
Title: Efficacy of Topical 95% Trichloroaceteic Acid in the Treatment of CIN 1 or Less After Low-grade Abnormality of Screening Test: A Randomized Controlled Trial
Brief Title: Efficacy of Topical 95% TCA in the Treatment of CIN 1 or Less After Low-grade Abnormality of Screening Test
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: I have found it is quite difficult to conduct the work without changing some detail in original protocol. So we would like to re-start the study again with some modification.
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 154/2566
Record Dates: First submitted 2023-09-29; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-08

CONDITIONS: CIN1; Trichloroacetic Acid
MeSH Terms: interventions — Trichloroacetic Acid; Acetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TCA plus acetic acid 1 (Experimental): No lesion group,
  Interventions: Drug: Trichloroacetic acid
- Acetic acid 1 (No Intervention): No lesion group, Applying acetic acid which normally used during colposcopic examination at transformation zone during colposcopic examination
- TCA plus acetic acid 2 (Experimental): Having lesion with normal pathologic examination
  Interventions: Drug: Trichloroacetic acid
- Acetic acid 2 (No Intervention): Having lesion with normal pathologic examination, Applying acetic acid which normally used during colposcopic examination at transformation zone and lesion during colposcopic examination
- TCA plus acetic acid 3 (Experimental): Having lesion with low-grade abnomality on pathologic examination,
  Interventions: Drug: Trichloroacetic acid
- Acetic acid 3 (No Intervention): Having lesion with low-grade abnomality on pathologic examination, Applying acetic acid which normally used during colposcopic examination at transformation zone and lesion during colposcopic examination

INTERVENTIONS:
Drug: Trichloroacetic acid — Applying Trichloroacetic acid 95 % topical solution plus acetic acid at the transformation zone or lesion (if have) of the cervix during colposcopic examination (95% topical trichloroacetic acid is used just before finishing examination, while acetic acid is used normally when perform colposcopy)
  Other Names: Trichloroacetic acid plus Acetic acid
  Arms: TCA plus acetic acid 1; TCA plus acetic acid 2; TCA plus acetic acid 3

SUMMARY:
To evaluate the efficacy of topical 95% TCA in the treatment of CIN 1 or less after low grade abnormality of screening test

DETAILED DESCRIPTION:
The patients meeting inclusion criteria were initially divided into two groups which are no lesion and having lesion at cervix on colposcopic examination.

Participant in no lesion group were divided into two group, recieving 95% Trichloroacetic acid (intervention) plus aceteic acid (commonly apply at cervix during colposcopic examination) applying to the cervix at T-zone and Acetic acid alone group.

We follow-up each group for 6 months to evaluate the outcome using cytologic examination, HPV testing and colposcopic examination (also biopsy if lesion is seen) compare to previous result (before treatment)

In the group having lesion at cervix, we initially biopsy the lesion and wait for pathologic result. If the pathologic results are high-grade lesion e.g. HSIL, we exclude them from this study. On the contrary, if the pathologic result s are low-grade lesion, we divided them into two group, normal pathologic exam and low-grade abnormality on pathologic examination. Both of them are divided into two groups and follow-up for 6 months, similar to the no lesion group

* During colposcopic examination, we also repeat cytologic examination and HPV testing as well

** Pregnancy test is done before applying 95%Trichloroacetic acid and at the time of follow-up. If positive at any point of time, participants are excluded from the study

ELIGIBILITY:
Inclusion Criteria:

* Women who have low-grade abnormality result such as ASC-US, LSIL, HPV 16/18 positive, persistent HPV infection after cervical cancer screening test
* No history of endometrial or cervical cancer
* Pregnancy test negative
* Good communication in Thai language
* Vouluntarily participate to the study

Exclusion Criteria:

* Pregnancy test positive after participate in the study
* Pathologic result from colposcopic biopsy (before intervention) is high-grade abnormality such as HSIL, CIN2-3 or AIS

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with cytologic examination, HPV testing and colposcopic examination with biopsy ( Efficacy of 95%Trichloroacetic acid in the treatment of CIN1 or less) | 6 months after intervention
  using cytologic examination, HPV testing and colposcopic examination with biopsy (if having lesion) compare to previous results
  If all of the test's results are normal, we consider it as remission of CIN1 or less
  *normal means: Cytologic examination = Negative for intraepithelial lesion or malignancy HPV testing = no HPV detected Colposcopic examination not seen any lesion = normal (not perform biopsy) Colposcopic examination with biopsy = normal pathlogic result

SECONDARY OUTCOMES:
Pain after treatment which evaluated by using visual analogue scale | immediately after intervention, up to 2 weeks after intervention
  Sides effect of 95%Trichloroacetic acid
Having leukorrhea or not? which is recorded by questionnaire | immediately after intervention, up to 2 weeks after intervention
  Sides effect of 95%Trichloroacetic acid
Having abnormal vaginal bleeding or not? which is recorded by questionnaire | immediately after intervention, up to 2 weeks after intervention
  Sides effect of 95%Trichloroacetic acid

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Phaya Thai, Bangkok, Thailand